CLINICAL TRIAL: NCT03117608
Title: A SINGLE-BLIND, RANDOMIZED, CONTROLLED STUDY OF A SINGLE, INTRA-ARTICULAR INJECTION OF AUTOLOGOUS MICRO-FRAGMENTED ADIPOSE TISSUE (aMAT) VERSUS (VS) PRP IN PATIENTS WITH OSTEOARTHRITIS (OA) OF THE KNEE
Brief Title: A Single Intra-articular Injection of aMAT vs PRP in Patients With OA of the Knee
Acronym: LIPOJOINT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lipogems International spa (Industry)
Responsible Party: Principal Investigator, Prof. Marcacci, Principal Investigator, Lipogems International spa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIPOJOINT
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis, Knee
Keywords: OA; aMAT; PRP
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AUTOLOGOUS MICRO-FRAGMENTED ADIPOSE TISSUE (aMAT) (Experimental): injection of aMAT obtained with Lipogems® technology.
  Interventions: Biological: injection of autologous micro-fragmented adipose tissue (aMAT)
- platelet-rich plasma (PRP) (Active Comparator): single injection of platelet-rich plasma
  Interventions: Biological: injection of Platelet-rich Plasma (PRP)

INTERVENTIONS:
Biological: injection of autologous micro-fragmented adipose tissue (aMAT) — adipose tissue will be obtained from abdominal region or buttocks and aMAT, and processed with Lipogems® technology.
  Arms: AUTOLOGOUS MICRO-FRAGMENTED ADIPOSE TISSUE (aMAT)
Biological: injection of Platelet-rich Plasma (PRP) — injection of platelet-rich plasma
  Arms: platelet-rich plasma (PRP)

SUMMARY:
The study proposes to compare performances and safety of intra-articular injections of aMAT with those of a control group (PRP injections) for the treatment of symptomatic OA of the knee. The end-points will be determined evaluating the performances of the treatment group in terms of improvement of the symptomatology, functional recovery and radiological appearance.

DETAILED DESCRIPTION:
The clinical trial is a prospective, randomized, controlled, two-arm, single-blind study, involving 118 patients affected by symptomatic OA of the knee joint. Eligible subjects will be randomly allocated to one of the two treatment groups, with a 1:1 randomization ratio. Respectively, 59 patients treated with a single intra-articular injection of aMAT, and 59 patients treated with a single intra-articular injection of PRP.

The patients enrolled in the study will be treated according to the study protocol and followed after treatment with periodic visits and diagnostic imaging examinations, as Magnetic Resonance Imaging at twelve and twenty-four months follow-up and X-Ray, at three, six, twelve, and twenty-four months of follow-up.

ELIGIBILITY:
Inclusion Criteria

1. Patients provided written informed consent;
2. Patients aged between 18 and 75 years;
3. Knee symptomatic OA (Kellgren-Lawrence grade 1-4)
4. Failure of conservative treatment for at least 3 months;
5. Patients agreed to actively participate in the rehabilitation protocol and follow-up program;
6. Male or female patients;
7. Women of childbearing age had to use a proven method to prevent pregnancy, before the surgical treatment.

Exclusion Criteria

1. Patients incapable to understanding and will;
2. Patients participating in previous, concurrent or not, trials (ongoing or completed within three months);
3. Patients surgically treated for the same defect within one year;
4. Patients affected by malignancy;
5. Patients affected by metabolic or thyroid disorders;
6. Patients used to alcohol or drug (medication) abuse;
7. Patients affected by synovitis;
8. Varus or valgus misalignment exceeding 15°;
9. Body Mass Index > 40;
10. Patients with trauma within 6 months pre-operative.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2017-02-24 (Actual); Primary Completion 2022-08-24 (Estimated); Study Completion 2024-02-24 (Estimated)

PRIMARY OUTCOMES:
Safety | Time Frame: 24 months evaluation
  Safety of the procedure, documenting characteristics and incidence of adverse events.(AE)
clinical improvement documented with IKDC(International Knee Documentation Committee) score and KOOS (Knee Injury and Osteoarthritis Outcome Score) | Time Frame: 6 months evaluation
  change in IKDC and KOOS score

SECONDARY OUTCOMES:
stability of the clinical improvement documented with International Knee Documentation Committee (IKDC) score | Time Frame: 6, 24 months evaluation
  Change in IKDC Subjective score from baseline to follow up
stability of the clinical improvement documented with Knee Injury and Osteoarthritis Outcome Score (KOOS) | Time Frame: 3,6, 12, 24 months evaluation
  Change in KOOS score from baseline to follow up

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Versari, Study Director — Lipogems International spa
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided